CLINICAL TRIAL: NCT04303936
Title: PHYSICAL ACTIVITY AND FVIII CLEARANCE: RELEVANCE FOR PERSONALIZED THERAPY IN SEVERE HAEMOPHILIA A
Brief Title: PHYSICAL ACTIVITY AND FVIII CLEARANCE: RELEVANCE FOR PERSONALIZED THERAPY IN SEVERE HAEMOPHILIA A (PHYSEMO)
Acronym: PHYSEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Raimondo De Cristofaro, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2364
Record Dates: First submitted 2020-01-16; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with severe HA under FVIII concentrates prophylaxis (Other)
  Interventions: Device: SenseWear® armband device

INTERVENTIONS:
Device: SenseWear® armband device — Metabolic Holter, Physical Activity and Lifestyle, Portable outpatient "multi-sensor" energy consumption in calories (EE), movement, physical activity, quality of life, sleep

SUMMARY:
In persons with severe haemophilia A (HA) infused factor VIII (FVIII) half-life and other pharmacokinetic parameters can vary according to determinants such as blood group, von Willebrand factor (VWF) level or age. However, FVIII pharmacokinetics (PK) has not been thoroughly studied in patients with severe HA as a function of daily physical activity.

Patients with severe HA (FVIII <1%) are predisposed to prolonged bleeding following even minimal musculoskeletal injuries. Potential consequences of repeated musculoskeletal bleeding are pain, arthropathy and physical disability. The key standard of care for HA patients is prophylactic infusions of FVIII concentrates (25-50 IU kg-1 infused 2-3 x/week), depending on individual response.

The level of infused FVIII decreases as a function of time according to both specific PK features of each product and biochemical/genetic characteristics of the patients or different clinical conditions.

Some critical points remain still unraveled, for instance, whether or not FVIII AUC is significantly affected by physical activity/exercise, in response to increased metabolic rate or subclinical/microhaemorrhages in patients with severe HA.

It is known that vigorous-intensity physical activity/exercise can transiently but significantly increase circulating levels of endogenous VWF and consequently FVIII in normal subjects and in patients with moderate or mild haemophilia A. The proposed study is a Proof of Concept one as it will be aimed at investigating the relation between daily physical activity, measured by SenseWear® armband device, as number of daily steps, and PK variability of infused rec-FVIII concentrate. This kind of investigation has never been done and it is a great interest also for the evaluation of patients' quality of life.

DETAILED DESCRIPTION:
Background In persons with severe haemophilia A (HA) infused factor VIII (FVIII) half-life and other pharmacokinetic parameters can vary according to determinants such as blood group, von Willebrand factor (VWF) level or age [1]. However, FVIII pharmacokinetics (PK) has not been thoroughly studied in patients with severe HA as a function of daily physical activity, reliably measured with multi-dimensional parameters. Research has indeed demonstrated the benefits of physical activity and the negative consequences of sedentary behavior for physical and mental wellbeing [2]. Thus, physical activity has become increasingly prominent as an intervention tool; however, research is often hindered by the challenge of employing a valid, reliable measure that also adequately satisfies the research question or design [2, 3]. Patients with severe HA (FVIII <1%) are predisposed to prolonged bleeding following even minimal musculoskeletal injuries. Potential consequences of repeated musculoskeletal bleeding are pain, arthropathy and physical disability [4, 5]. The key standard of care for HA patients is prophylactic infusions of FVIII concentrates. Commonly used prophylaxis regimens with standard FVIII concentrates are 25-50 IU kg-1 infused 2-3 x/week, depending on individual response and/or resource availability of therapeutical products [6]. International guidelines also recommend to increase FVIII levels following musculoskeletal or other bleeds [6]. The level of infused FVIII decreases as a function of time according to both specific PK features of each product and biochemical/genetic characteristics of the patients or different clinical conditions. FVIII half-life is approximately 8-12 h [6]. FVIII half-life is increased in adult vs. pediatric patients [7, 8], in subjects with higher baseline von Willebrand factor (VWF) plasma levels [9, 10] and is decreased in patients with blood group O [8, 9]. On the other hand, some critical points remain still unraveled. One may wonder, for instance, whether or not FVIII AUC is significantly affected by physical activity/exercise, in response to increased metabolic rate or subclinical/microhaemorrhages in patients with severe HA [11]. It is known that vigorous-intensity physical activity/exercise can transiently but significantly increase circulating levels of endogenous VWF and consequently FVIII in normal subjects [12, 13]and in patients with moderate or mild haemophilia A [14, 15]. The proposed study is a Proof of Concept one as it will be aimed at investigating the relation between daily physical activity, measured by SenseWear® armband device, as number of daily steps, and PK variability of infused rec-FVIII concentrate. This kind of investigation has never been done and it is a great interest also for the evaluation of patients' quality of life.

Study design

This is a prospective, interventional, low risk, cohort study with device. Twenty patients (haemophilia A is a rare disease, hence the investigators are going to enroll in the study all the available patients), all consecutively enrolled in a period of 12 months, in the two, mentioned above, participant centers, will be followed for 12 months from the enrolment. Hence, the planned study period is as follows:

* initiation Q1 2019
* completion Q3 2020 Eligible patients will be asked not to use FVIII during the 72 hours before their baseline visit for the assessment of FVIII PK parameters. Two days before their visit to the clinic, patients will be asked to complete a questionnaire to give information on their general health status and use of medication in the preceding days. At baseline, T=0, following the routine clinical practice in the follow up of haemophilic patients, blood samples will be collected by venipuncture into plastic tubes containing 0.109 M buffered trisodium citrate in a 9:1 ratio. Blood sample will be taken and FVIII PK parameters will be determined and the SenseWear™ Armband will be put on place. Then, 50 IU/kg of the FVIII product, regularly used by the patient, will be infused. After infusion with FVIII, blood samples will be collected at 30 minutes and 1, 8, 24, 48 and 72 hours. The blood samples will be centrifuged for 15 minutes at 1500 × g (3000 rpm) immediately and plasma will be stored at -80°C.Patients will wear the SenseWear™ Armbandfor 7 consecutive days for at least 20 h/day.

A questionnaire on the quality of life (Haem-A-QoL)[17] will be administered to all enrolled patients (see Annex 3), following the routine clinical practice.

Methods Coagulation and haematology assays All hemostasis-related tests will be performed at the Hemostasis and Thrombosis Center of FPG. FVIII activity will be determined using the one-stage method. Since inhibitory antibodies against factor VIII may influence FVIII half-life, the presence of these antibodies will be assessed in pre-infusion samples using the Nijmegen variant of the Bethesda assay [16]. Inhibitor concentrations of >0.6 Bethesda Units (BU)/mL will be considered positive. Pre-infusion von Willebrand factor (VWF) antigen and activity levels will be determined using an immunometric assay (VWF:Ag and VWF:act) on an automatic chemiluminescence instrument (AcuStar, Instrumentation Laboratory, Werfen Group, Milano, Italy).

Method to measure physical activity of patients Physical activity will be measured using the SenseWear™ Armband (see the enclosed file for the description of the device's characteristics, Annex 2) and the balanced daily energy expenditure, number of steps, physical activity intensity (METs) will be monitored for each subject in the period of observation. The device is worn over the right triceps brachii muscle and incorporates five sensors: two-axis accelerometer (for movement patterns and step-count), galvanic skin response, skin temperature, near body temperature sensor and heat flux [1]. According to the study protocol, patients will wear the SenseWear™ Armband on 7 consecutive days for at least 20 h/day. Collected data will be exported via the Professional InnerView Software 7.0 (Body Media Inc., Pittsburgh, PA). This software calculates the balanced daily energy expenditure (EE) from the sensor parameters together with anthropometric data (gender, age, height, weight, BMI, handedness, smoking status). Physical activity intensity is classified by Metabolic Equivalents of Task (MET) as defined by Jette et al. [2], which are commonly used to classify activities based on their EE.

Physical Examinations At screening and subsequent study visits a physical examination will be performed on the following body systems being described as normal or abnormal: general appearance, headand neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological. At screening, if an abnormal condition is detected, the condition will be described on the medical history CRF. At study visit, if a new abnormal or worsened abnormal pre-existing condition is detected, the condition will be described on the CRF.

Vital Signs Vital signs will include height (cm) and weight (kg). Height and weight will be collected,if available, at screening visit and study completion/termination.

Subject Identification Code The following series of numbers will comprise the subject identification code (SIC): protocol acronym (PHYSEMO), and 2-digit subject number (e.g., 01….02) reflecting the order of enrollment (i.e., signing the informed consent form). For example, the third subject who signed an informed consent form will be identified as PHYSEMO-03. All study documents (e.g., CRFs, clinical documentation, etc.) will be identified with the SIC.

Subject completation/discontinuation Reasons for completion/discontinuation will be reported on the Completion/ Discontinuation CRF page, including: completed, screen failure, adverse event (e.g., death), discontinuation by subject (e.g., lost to follow-up[defined as 3 documented unsuccessful attempts to contact the subject], dropout),physician decision (e.g., pregnancy, progressive disease, protocol violation(s)). Regardless of the reason, all data available for the subject up to the time of completion/ discontinuation should be recorded on the appropriate CRF pages. The reason for discontinuation will be recorded on the CRF, and data collected up to the time of discontinuation will be used in the analysis and included in the clinical study report.

Procedures for Monitoring Subject Compliance There is no procedure for monitoring subject compliance. All treatment regimens and monitoring schedules will be determined by the treating physician. The protocol does not require for any additional testing or monitoring than what is judged necessary by the treating physician.

Statistics and data analysis Major baseline demographic, anthropometric and clinical variables will be summarized for the enrolled populations. All continuous variables will be summarized with means, standard deviations, medians, interquartile ranges, minimums, and maximums. Categorical variables will be summarized with frequencies and percentages. Age, body mass index, annual bleeding rate (ABR) and Hemophilia Joint Heath Score (HJHS) score will be registered at the enrollment visit according to routine good clinical practice for heamophilia patients and described statistically. In order to investigate whether the daily physical activity level affects the PK parameter: AUC, the correctness of the experience of clinicians, which suggests a higher level of physical activity in the 12-35 age group, will be demonstrated first. Later the investigators will demonstrate that the mean AUC of the 12-35 group is significantly smaller than the mean AUC of the 36-60 group, using the appropriate test according to the variables' nature. This strategy will allow to analyze the influence of physical activity inside each group on PK parameters of patients with more homogeneous characteristics.

Linear regression analysis (bivariate, Spearman method) will be used to assess the relation between FVIII PK parameters and several independent variables, such as age, known blood group, VWF antigen/activity, physical activity parameters measured using the SenseWear™ Armband and HJHS score. Furthermore, since the HJHS scores are dependent on age [18, 19], the findings will be adjusted for age at HJHS score. The independent variables that will be significantly associated with PK parameters (especially half-life and clearance) with p<0.05 will be analyzed in a multivariable analysis. The validated program MyPK Fit (Shire) will be used to calculate FVIII PK parameters. The last five years of follow-up will be used to estimate annual clotting factor use (IU/kg/yr), number of joint bleeds per year and weekly dose on prophylaxis (IU/kg/wk).

All the tests will be performed considering a level of confidence alpha=0.05. Analyses will be performed using SPSS software (version 21, Chicago, IL, USA) and GraphPad Prism software (GraphPad Software, Inc, La Jolla, CA, USA).

Sample Size Calculation Dealing with a rare disease and considering the amount of eligible patients available from both the centres, the expected sample size is roughly N=20 patients. A significant difference in daily physical activity level of at least 2000 steps was defined as the primary end-point and the level of physical activity corresponding to 6000 ± 2000 and 12000 ± 1000 steps was assumed for 36-60 and 12-35 years groups, respectively. A sample size of 10 subjects in each group was estimated for 80% power and alfa 0.05.

Handling of Missing, Unused, and Spurious Data Analyses will exclude missing data. Unused and spurious data will be listed in the Clinical Study Report to include the reason(s).

Ethics Committee and Regulatory Authorities Before enrollment of patients into this study, the protocol, informed consent form (see Annex 3), any promotional material/advertisements, and any other written information to be provided will be reviewed and approved/given favorable opinion by the EC and applicable regulatory authorities.

If the protocol or any other information given to the subject is amended, the revised documents will be reviewed and approved/given favorable opinion by the EC and applicable regulatory authorities, where applicable. The protocol amendment will only be implemented upon the sponsor's receipt of approval and, if required, upon the sponsor's notification of applicable regulatory authority(ies) approval.

Informed Consent Investigators will choose patients for enrollment based on the study eligibility criteria.

The investigator will exercise no selectivity so that no bias is introduced from this source.

All patients must sign an informed consent form before entering into the study according to applicable regulatory requirements. Before use, the informed consent form will be reviewed by the EC. The informed consent form will include a comprehensive explanation of the proposed treatment without any exculpatory statements. Patients will be allowed sufficient time to consider participation in the study. By signing the informed consent form, patients agree to take part in the study.

Confidentiality Policy The investigator will comply with the confidentiality policy as described in the Non-Interventional Trial Agreement.

Study Documents and Case Report Forms The investigator will maintain complete and accurate study documentation in a separate file. Documentation may include medical records, records detailing the progress of the study for each subject, signed informed consent forms, correspondence with the EC, enrollment and screening information, CRFs and laboratory reports. The investigator will comply with the procedures for data recording and reporting. Any corrections to study documentation must be performed as follows: 1) the first entry will be crossed out entirely, remaining legible; and 2) each correction must be dated and initialed by the person correcting the entry; the use of correction fluid and erasing are prohibited.

Case Report Forms The investigator is responsible for the procurement of data and for the quality of data recorded on the CRFs. CRFs will be provided in paper form.

Only authorized study site personnel will record or change data on the CRFs. All data should preferably be entered on the CRFs during the study visit. Changes to a CRF will require documentation of the reason for each change.

The handling of data by the sponsor, including data quality assurance, will comply with regulatory guidelines and the standard operating procedures of the sponsor. Data management and control processes specific to the study will be described in the data management plan.

Document and Data Retention The investigator will retain study documentation and data in accordance with applicable regulatory requirements and the document and data retention policy, as described in the Non-Interventional Study Agreement.

ELIGIBILITY:
Inclusion Criteria:

* Patients (12-60 yr. old) with severe HA under FVIII concentrates prophylaxis will be selected at the Haemostasis and Thrombosis Center of the Fondazione Policlinico Universitario "A. Gemelli", IRCCS, Rome, Italy (FPG) and at the satellite site at the Department of Cellular Biotechnology and Haemathology, Policlinico Umberto I, Sapienza University of Rome, Italy (UNSA_SS).

Exclusion Criteria:

* All patients with malignant tumors, or treated with anticoagulant / antiplatelet agents, and suffering from other congenital coagulation disorders (von disease Willebrand disease, other congenital deficiency of coagulation factors) or severe thrombocytopenia (<30,000 Plt /μL).

Patients who would have undergone a severe bleed or surgery during the past 3 months before enrolment.

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Study of the association between physical activity, measured by mean number of daily steps, with the Area Under the Curve (AUC) PK parameter in patients with severe HA under prophylaxis. | 12 months
  Investigate whether and how the daily physical activity (measured as number of steps, using the SenseWear™ Armband device) affects the PK parameter. In more details, the study aims to evaluate whether and how the FVIII AUC PK parameter is significantly associated with the mean number of daily steps in patients with severe HA.

SECONDARY OUTCOMES:
Study of the association between physical activity, measured by the mean number of daily steps, with the clearance (U/ml/hr) of FVIII concentrate PK parameters in patients with severe HA. | 12 months
  Investigate whether and how the daily physical activity (measured as mean number of daily steps, using the SenseWear™ Armband device) affects the PK parameter. In more details, the study aims to evaluate whether and how the FVIII clearance (U/ml/hr) PK parameter is significantly associated with the number of steps in patients with severe HA.
Study of the association between physical activity, measured by the mean number of daily steps, with half life (hr) of FVIII concentrate PK parameters in patients with severe HA. | 12 months
  Investigate whether and how the daily physical activity (measured as mean number of daily steps, using the SenseWear™ Armband device) affects the PK parameter. In more details, the study aims to evaluate whether and how the half life (hr) PK parameter is significantly associated with the number of steps in patients with severe HA.
Physical activity (mean number of daily steps) level and HJHS score | 12 months
  To assess whether and how the physical activity (measured by mean number of daily steps), measured by the SenseWear™ Armband device, is significantly associated with the HJHS score;
Physical activity, measured by mean number of daily steps, andHaem-A-QoL score | 12 months
  To assess whether and how the physical activity, measured by mean number of daily steps) using the SenseWear™ Armband device, is significantly associated with the Haem-A-QoL score.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kepa S, Horvath B, Reitter-Pfoertner S, Schemper M, Quehenberger P, Grundbichler M, Heistinger M, Neumeister P, Mannhalter C, Pabinger I. Parameters influencing FVIII pharmacokinetics in patients with severe and moderate haemophilia A. Haemophilia. 2015 May;21(3):343-350. doi: 10.1111/hae.12592. Epub 2015 Jan 13. PMID 25582282
- [Background] Lee IM, Hsieh CC, Paffenbarger RS Jr. Exercise intensity and longevity in men. The Harvard Alumni Health Study. JAMA. 1995 Apr 19;273(15):1179-84. PMID 7707624
- [Background] Macfarlane DJ, Lee CC, Ho EY, Chan KL, Chan D. Convergent validity of six methods to assess physical activity in daily life. J Appl Physiol (1985). 2006 Nov;101(5):1328-34. doi: 10.1152/japplphysiol.00336.2006. Epub 2006 Jul 6. PMID 16825525
- [Background] Hoots WK, Rodriguez N, Boggio L, Valentino LA. Pathogenesis of haemophilic synovitis: clinical aspects. Haemophilia. 2007 Nov;13 Suppl 3:4-9. doi: 10.1111/j.1365-2516.2007.01533.x. PMID 17822514
- [Background] Lafeber FP, Miossec P, Valentino LA. Physiopathology of haemophilic arthropathy. Haemophilia. 2008 Jul;14 Suppl 4:3-9. doi: 10.1111/j.1365-2516.2008.01732.x. PMID 18494686
- [Background] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Background] Blanchette VS, Shapiro AD, Liesner RJ, Hernandez Navarro F, Warrier I, Schroth PC, Spotts G, Ewenstein BM; rAHF-PFM Clinical Study Group. Plasma and albumin-free recombinant factor VIII: pharmacokinetics, efficacy and safety in previously treated pediatric patients. J Thromb Haemost. 2008 Aug;6(8):1319-26. doi: 10.1111/j.1538-7836.2008.03032.x. Epub 2008 May 22. PMID 18503631
- [Background] Collins PW, Bjorkman S, Fischer K, Blanchette V, Oh M, Schroth P, Fritsch S, Casey K, Spotts G, Ewenstein BM. Factor VIII requirement to maintain a target plasma level in the prophylactic treatment of severe hemophilia A: influences of variance in pharmacokinetics and treatment regimens. J Thromb Haemost. 2010 Feb;8(2):269-75. doi: 10.1111/j.1538-7836.2009.03703.x. Epub 2009 Nov 23. PMID 19943875
- [Background] van Dijk K, van der Bom JG, Lenting PJ, de Groot PG, Mauser-Bunschoten EP, Roosendaal G, Grobbee DE, van den Berg HM. Factor VIII half-life and clinical phenotype of severe hemophilia A. Haematologica. 2005 Apr;90(4):494-8. PMID 15820945
- [Background] Lalezari S, Martinowitz U, Windyga J, Enriquez MM, Delesen H, Schwartz L, Scharrer I. Correlation between endogenous VWF:Ag and PK parameters and bleeding frequency in severe haemophilia A subjects during three-times-weekly prophylaxis with rFVIII-FS. Haemophilia. 2014 Jan;20(1):e15-22. doi: 10.1111/hae.12294. Epub 2013 Nov 20. PMID 24252058
- [Background] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Background] Smith JE. Effects of strenuous exercise on haemostasis. Br J Sports Med. 2003;37(5):433-5. doi: 10.1136/bjsm.37.5.433. PMID 14514536
- [Background] Lippi G, Maffulli N. Biological influence of physical exercise on hemostasis. Semin Thromb Hemost. 2009 Apr;35(3):269-76. doi: 10.1055/s-0029-1222605. Epub 2009 May 18. PMID 19452402
- [Background] Groen WG, den Uijl IE, van der Net J, Grobbee DE, de Groot PG, Fischer K. Protected by nature? Effects of strenuous physical exercise on FVIII activity in moderate and mild haemophilia A patients: a pilot study. Haemophilia. 2013 Jul;19(4):519-23. doi: 10.1111/hae.12111. Epub 2013 Mar 19. PMID 23510308
- [Background] Zourikian N, Merlen C, Bonnefoy A, St-Louis J, Rivard GE. Effects of moderate-intensity physical exercise on pharmacokinetics of factor VIII and von Willebrand factor in young adults with severe haemophilia A: a pilot study. Haemophilia. 2016 May;22(3):e177-83. doi: 10.1111/hae.12869. Epub 2016 Mar 14. PMID 26988074
- [Background] Arranz P, Remor E, Quintana M, Villar A, Diaz JL, Moreno M, Monteagudo J, Ugarriza A, Soto I, Perez R, Chacon J, Garcia-Luaces M, Cid A, Balda I, Lopez MF, Gutierrez MJ, Martinez E, Marrero C, Prieto M, Sedano C, Vaca R, Altisent C, Hernandez-Navarro F; Hemofilia-QoL Group. Development of a new disease-specific quality-of-life questionnaire to adults living with haemophilia. Haemophilia. 2004 Jul;10(4):376-82. doi: 10.1111/j.1365-2516.2004.00918.x. PMID 15230953
- [Background] Chang CY, Li TY, Cheng SN, Pan RY, Wang HJ, Lin SY, Chen YC. Prevalence and severity by age and other clinical correlates of haemophilic arthropathy of the elbow, knee and ankle among Taiwanese patients with haemophilia. Haemophilia. 2017 Mar;23(2):284-291. doi: 10.1111/hae.13117. Epub 2016 Nov 8. PMID 27862662